CLINICAL TRIAL: NCT05043896
Title: The Effect of Combination Therapy Using Li-ESWT (Low Intensity Extracorporeal Shockwave Therapy) and PDE-5 Inhibitor in Patients With Erectile Dysfunction
Brief Title: The Effect of Combination Therapy Using Li-ESWT and PDE-5 Inhibitor in Patients With Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Principal Investigator, Andrian, dr., Sp.And, Resident of Andrology Department, Principal Investigator, Medical Doctor, Dr. Soetomo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1690/KEPK/XII/2019
Record Dates: First submitted 2021-08-26; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Extracorporeal Shockwave Therapy; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination therapy (Experimental): Li-ESWT + tadalafil
  Interventions: Procedure: Li-ESWT; Drug: Tadalafil 2.5Mg Tab
- Single Therapy (Sham Comparator): tadalafil only
  Interventions: Drug: Tadalafil 2.5Mg Tab

INTERVENTIONS:
Procedure: Li-ESWT — Li-ESWT twice weekly for 4 weeks
  Other Names: Shockwave Therapy
  Arms: Combination therapy
Drug: Tadalafil 2.5Mg Tab — tadalafil 2.5mg once daily
  Other Names: Standard First Line Therapy

SUMMARY:
to compare the effect of combination of li-eswt and pde-5 inhibitor to pde-5 alone in erectile dysfunction patients

DETAILED DESCRIPTION:
Comparing the effect of Combination therapy (Li-ESWT combined with PDE5-inhibitor) vs SIngle therapy (PDE5-inhibitor) in mild to moderate Erectile Dysfunction patients.

Parameters used for comparation are EHS score, IIEF-5 score, VEGF level and PSV

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate Erectile dysfunction
* Married
* Sexually active
* Consenting to participate in the trial

Exclusion Criteria:

* Psychological problems
* Spinal injury
* History of malignancy
* Penile anatomy abnormalities
* Allergic and Contraindications to tadalafil
* On anti-mitotic drugs

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only for male
Enrollment: 30 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Erectile Hardness Score (EHS) | 4 weeks
  Developed in 1998, the EHS is a single-item Likert scale that men can use on their own.
  The tool asks them to consider the question "How would you rate the hardness of your erection?" and select one of the following options:
  0 Penis does not enlarge
  1. Penis is larger, but not hard
  2. Penis is hard, but not hard enough for penetration
  3. Penis is hard enough for penetration, but not completely hard
  4. Penis is completely hard and fully rigid
  The EHS score was taken pre and post intervention
International Index of Erectile Function (IIEF-5) score | 4 weeks
  IIEF-5 is a tool for ED (Erectile Dysfunction)diagnosis. The possible scores for the IIEF-5 range from 5 to 25, and ED was classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25)
  IIEF-5 score was taken pre and post intervention
Peak Systolic Velocity (PSV) | 4 weeks
  PSV was measured in cm/s, by using Doppler Ultrasonography. The probe is located at the penis, to be precise in the penoscrotal junction, to measure the velocity of the blood flow in the cavernous arteries.
  The test was done in flaccid state of the penis Measurement was taken by an experienced ultrasonographer in the radiology unit. Measurement was taken pre and post intervention
Vascular Endothelial Growth Factor (VEGF) level in plasma | 4 weeks
  VEGF was measured in pg/ml. VEGF test were done by blood test in the laboratory using the VEGF-A ELISA Kit.
  Blood for tests were drawn pre and post test

CONTACTS AND LOCATIONS:
Overall Officials: Tjahjo Tanojo, dr, Principal Investigator — Dr. Soetomo General Hospital, Andrology Clinic
Locations (1):
- dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (5):
  • Study Protocol: Study Protocol Chart (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT05043896/Prot_000.pdf
  • Study Protocol: Ethical Clearance (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT05043896/Prot_001.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocols and Statistical Analysis Plan (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT05043896/Prot_SAP_002.pdf
  • Statistical Analysis Plan: Statistics Results (2020-06-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT05043896/SAP_003.pdf
  • Informed Consent Form (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT05043896/ICF_004.pdf